CLINICAL TRIAL: NCT03515070
Title: Microbiome and Genetic Analysis of Family Members With Inflammatory Bowel Disease
Brief Title: Microbiome and Genetic Analysis of Familial IBD
Status: Completed | Type: Observational
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Chang Kyun Lee, Professor, Kyunghee University Medical Center
Other Study IDs: Familial_IBD_Microbiome
Record Dates: First submitted 2018-04-22; First posted 2018-05-03 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Gastrointestinal Microbiome; Genetics
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and fecal sample from each study subjects
  * DNA extraction will be performed soon after the blood sampling.
  * Fecal sample will be prepped for the microbiome analysis and microbial 16 S RNA will be extracted from the sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel disease(IBD) is a chronic inflammatory condition for gastrointestinal tract.

Regarding its pathogenesis, there has been numerous studies to reveal the complex association between genetic and environmental factors.

In Korea, the incidence of IBD is growing rapidly but genetic studies solely including patients with Korean descent were not sufficient enough.

Therefore, the investigators planned to conduct genetic and fecal microbial analysis for the 60 individuals from 30 Korean IBD families to find out the pathogenesis of IBD.

DETAILED DESCRIPTION:
Under the hypothesis that more risk variants will be observed among the familial IBD patient than in IBD patients without any other affected family members, the investigators designed genetic and fecal microbiome analysis for 60 patients form 30 families.

After extracting the DNA from blood samples, whole genome sequencing will be performed and data will be comprared with the previously reported variances. Novel variances or incidence of specific variances will be measured.

Genome-wide single nucleotide polymorphism array using Immunochip will be performed to search common genetic variants and to calculate genetic risk score of IBD.

In this study, fecal microbiome is a surrogate marker for the enviromental aspect of pathogenesis of IBD. The investigators assumed that family members are sharing similar mode of lifestyle therefore we're presumed that their fecal microbial composition is alike.

Comparing genetic and microbial datas altogether with the data from unaffected family member(Healthy internal control), investigators expecting to explain the genetic and enviromental aspect of IBD pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* 60 individuals from 30 families of Crohn's disease or ulcerative colitis.
* Unaffected 30 individuals from each family as healthy internal control.

Exclusion Criteria:

* Person with history of using antibiotics or probiotics within previous 4 weeks.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators are planned to study family members with IBD(Crohn's disease or ulcerative colitis).
  They are all Koreal descent and study candidates are two patients from each 30 families. As a healthy internal control, another family member without IBD history will be also enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Rare genetic variants of inflammatory bowel disease | Three months after the sample collection
  Results from whole genome sequencing of blood samples of study participants. Planned to compare with the previously reported variances.
Common genetic variants of inflammatory bowel disease | Three months after the sample collection
  Results from genome-wide single nucleotide polymorphism array of blood samples of study participants.
  Planned to compare with the previously reported variances.
Genetic risk score of inflammatory bowel disease | Three months after the sample collection
  Results from genome-wide single nucleotide polymorphism array of blood samples of study participants.
  Planned to compare with the previously reported variances.
Fecal microbiome composition of each study subjects | Three months after the sample collection
  Microbial diversity measured from 16S RNA sequencing datas of fecal microbiomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Jong Kim, M.D. PhD, Principal Investigator — Kyung Hee University Hospital; Chang Kyun Lee, M.D. PhD, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
After publishing the results, any data sharing request from other researchers will be positively considered.
  But extent of sharing is not decided yet.

REFERENCES:
- [Background] Wellcome Trust Case Control Consortium. Genome-wide association study of 14,000 cases of seven common diseases and 3,000 shared controls. Nature. 2007 Jun 7;447(7145):661-78. doi: 10.1038/nature05911. PMID 17554300
- [Background] Thia KT, Loftus EV Jr, Sandborn WJ, Yang SK. An update on the epidemiology of inflammatory bowel disease in Asia. Am J Gastroenterol. 2008 Dec;103(12):3167-82. doi: 10.1111/j.1572-0241.2008.02158.x. PMID 19086963
- [Background] Lashner BA, Evans AA, Kirsner JB, Hanauer SB. Prevalence and incidence of inflammatory bowel disease in family members. Gastroenterology. 1986 Dec;91(6):1396-400. doi: 10.1016/0016-5085(86)90193-9. PMID 3770366
- [Background] Stittrich AB, Ashworth J, Shi M, Robinson M, Mauldin D, Brunkow ME, Biswas S, Kim JM, Kwon KS, Jung JU, Galas D, Serikawa K, Duerr RH, Guthery SL, Peschon J, Hood L, Roach JC, Glusman G. Genomic architecture of inflammatory bowel disease in five families with multiple affected individuals. Hum Genome Var. 2016 Jan 7;3:15060. doi: 10.1038/hgv.2015.60. eCollection 2016. PMID 27081563
- [Background] Jostins L, Ripke S, Weersma RK, Duerr RH, McGovern DP, Hui KY, Lee JC, Schumm LP, Sharma Y, Anderson CA, Essers J, Mitrovic M, Ning K, Cleynen I, Theatre E, Spain SL, Raychaudhuri S, Goyette P, Wei Z, Abraham C, Achkar JP, Ahmad T, Amininejad L, Ananthakrishnan AN, Andersen V, Andrews JM, Baidoo L, Balschun T, Bampton PA, Bitton A, Boucher G, Brand S, Buning C, Cohain A, Cichon S, D'Amato M, De Jong D, Devaney KL, Dubinsky M, Edwards C, Ellinghaus D, Ferguson LR, Franchimont D, Fransen K, Gearry R, Georges M, Gieger C, Glas J, Haritunians T, Hart A, Hawkey C, Hedl M, Hu X, Karlsen TH, Kupcinskas L, Kugathasan S, Latiano A, Laukens D, Lawrance IC, Lees CW, Louis E, Mahy G, Mansfield J, Morgan AR, Mowat C, Newman W, Palmieri O, Ponsioen CY, Potocnik U, Prescott NJ, Regueiro M, Rotter JI, Russell RK, Sanderson JD, Sans M, Satsangi J, Schreiber S, Simms LA, Sventoraityte J, Targan SR, Taylor KD, Tremelling M, Verspaget HW, De Vos M, Wijmenga C, Wilson DC, Winkelmann J, Xavier RJ, Zeissig S, Zhang B, Zhang CK, Zhao H; International IBD Genetics Consortium (IIBDGC); Silverberg MS, Annese V, Hakonarson H, Brant SR, Radford-Smith G, Mathew CG, Rioux JD, Schadt EE, Daly MJ, Franke A, Parkes M, Vermeire S, Barrett JC, Cho JH. Host-microbe interactions have shaped the genetic architecture of inflammatory bowel disease. Nature. 2012 Nov 1;491(7422):119-24. doi: 10.1038/nature11582. PMID 23128233